CLINICAL TRIAL: NCT03535441
Title: Evidence for SIRT1 Mediated HMGB1 Release From Kidney Cells in the Early Stages of Hemorrhagic Shock
Brief Title: HMGB1 Release From Hemorrhagic Shock Patients
Status: Completed | Type: Observational
Sponsor: Xingui Dai (Other)
Responsible Party: Sponsor-Investigator, Xingui Dai, serum HHMGB1 concentration of hemorrhagic shock patients, First People's Hospital of Chenzhou
Organization: First People's Hospital of Chenzhou (Other)
Other Study IDs: HSHMGB12018
Record Dates: First submitted 2018-05-11; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Intensive Care Unit; Hemorrhagic Shock; Adult Disease
Keywords: hemorrhagic shock; HMGB1
MeSH Terms: conditions — Shock, Hemorrhagic; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- voluteer group: No treatment, only blood sample collection
- hemorrhagic shock group: HS was defined as out-of-hospital systolic blood pressure (SBP) of 70 mmHg or less or SBP ranging 71 to 90 mmHg with a heart rate of 108 beats/min or more. Exclusion criteria were pregnancy, <15 years old, more than 2,000 mL of intravenous fluids or blood before enrollment, hypothermia, drowning, asphyxia, burns, isolated penetrating head injury, time of call received by dispatch to study intervention longer than 4 h, known prisoners, and transfer from another hospital

SUMMARY:
It is reported that high mobility group box 1 (HMGB1), a non-histone nuclear protein, can serve as an alarmin with damage associated molecular patterns to activate immune responses in the early stages of hemorrhagic shock (HS). However, the origin of HMGB1 and how it is released following HS is poorly understood. In this study, we teased out this mechanism. We try to record the concentration of serum HMGB1 protein following HS in clinical patients.

DETAILED DESCRIPTION:
The study was approved by the First People's Hospital of Chenzhou, Hunan, P.R. China. Consent was obtained from patients in their hospital course. Eighteen patients were enrolled for each group. In addition, Acute Physiological and Chronic Health Evaluation II (APACHE II) score was used to evaluate the severity and morbidity of HS patients Serial blood samples were collected at indicated time points on hospital admission for HS patients (0, 2, 4, 8, 24, and 72 h following HS). Levels of HMGB1 were detected by ELISA according to the kit manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

Hemorrhagic shock (HS) was defined as out-of-hospital systolic blood pressure (SBP) of 70 mmHg or less or SBP ranging 71 to 90 mmHg with a heart rate of 108 beats/min or more.

Exclusion Criteria:

pregnancy, <18 years old, more than 2,000 mL of intravenous fluids or blood before enrollment, hypothermia, drowning, asphyxia, burns, isolated penetrating head injury, time of call received by dispatch to study intervention longer than 4 h, known prisoners, and transfer from another hospital

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers OR Hemorrhagic shock (HS) patients enrolled in ICU
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
serum HMGB1 concentration | 24 hours following hemorrhagic shock
  the concentration of serum HMGB1 were progressively increased following Hemorrhagic shock

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Chenzhou, Chenzhou, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Hemorrhagic shock (HS) is a pathologic process caused by insufficient perfusion in multiple organs, and usually initiates a systemic post-traumatic inflammation response. The resulting increased inflammation response may accelerate the multiple organ dysfunctions . Extracellular high-mobility group box 1 (HMGB1) was found to mediate inflammation during sterile and infectious injury and contributes significantly to disease pathogenesis. However, the exact role of HMGB1-mediated inflammation in HS is not fully understood.
  In this study, we first test the serum HMGB1 concentration in clinical HS patients and then we explored the underlying mechanism in HS animal model. An unexpected mechanism of HMGB1 released from multiple organs (especially in kidney) was found.
Time Frame: 72 hours following hemorrhagic shock
Access Criteria: HS was defined as out-of-hospital systolic blood pressure (SBP) of 70 mmHg or less or SBP ranging 71 to 90 mmHg with a heart rate of 108 beats/min or more. Exclusion criteria were pregnancy, <18 years old, more than 2,000 mL of intravenous fluids or blood before enrollment, hypothermia, drowning, asphyxia, burns, isolated penetrating head injury, time of call received by dispatch to study intervention longer than 4 h, known prisoners, and transfer from another hospital

REFERENCES:
- [Result] Rickenbacher A, Jang JH, Limani P, Ungethum U, Lehmann K, Oberkofler CE, Weber A, Graf R, Humar B, Clavien PA. Fasting protects liver from ischemic injury through Sirt1-mediated downregulation of circulating HMGB1 in mice. J Hepatol. 2014 Aug;61(2):301-8. doi: 10.1016/j.jhep.2014.04.010. Epub 2014 Apr 18. PMID 24751831
- [Result] Rabadi MM, Xavier S, Vasko R, Kaur K, Goligorksy MS, Ratliff BB. High-mobility group box 1 is a novel deacetylation target of Sirtuin1. Kidney Int. 2015 Jan;87(1):95-108. doi: 10.1038/ki.2014.217. Epub 2014 Jun 18. PMID 24940804
- [Result] Hwang JS, Lee WJ, Kang ES, Ham SA, Yoo T, Paek KS, Lim DS, Do JT, Seo HG. Ligand-activated peroxisome proliferator-activated receptor-delta and -gamma inhibit lipopolysaccharide-primed release of high mobility group box 1 through upregulation of SIRT1. Cell Death Dis. 2014 Oct 2;5(10):e1432. doi: 10.1038/cddis.2014.406. PMID 25275593
- [Result] Hwang JS, Choi HS, Ham SA, Yoo T, Lee WJ, Paek KS, Seo HG. Deacetylation-mediated interaction of SIRT1-HMGB1 improves survival in a mouse model of endotoxemia. Sci Rep. 2015 Nov 2;5:15971. doi: 10.1038/srep15971. PMID 26522327